CLINICAL TRIAL: NCT02788929
Title: INCreasing Exercise adhereNce After percuTaneous Coronary InterVEntion With the Fitbit Charge HR Device: the INCENTIVE Trial
Brief Title: Increasing Exercise Adherence After Percutaneous Coronary Intervention With the Fitbit Charge HR Device
Acronym: INCENTIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Director of Cardiac Catheterization Laboratories, Professor of Medicine, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-008
Record Dates: First submitted 2016-05-20; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Acute Coronary Syndrome
Keywords: Percutaneous Transluminal Coronary Intervention; Cardiac Rehabilitation; Fitbit Charge HR
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fitbit Charge HR (Active Comparator): Use of the Fitbit Charge HR, a simple, user-friendly, wrist-worn, commercially available device which provides feedback on exercise goal adherence, in combination with the Fitbit mobile platform application.
  All patients will wear the Actigraph wGT3X-BT, from which data is extracted. Actigraph does not provide patient any feedback.
  Interventions: Device: Fitbit Charge HR
- No Device (No Intervention): No Fitbit used and no feedback on exercise goal adherence. All patients will wear the Actigraph wGT3X-BT, from which data is extracted. Actigraph does not provide patient any feedback.

INTERVENTIONS:
Device: Fitbit Charge HR — Patients randomized to the FitBit group will receive Fitbit Charge HR, a simple, user-friendly, wrist-worn, commercially available device which provides feedback on exercise goal adherence, in combination with the Fitbit mobile platform application.
  Arms: Fitbit Charge HR

SUMMARY:
Design: Single center, prospective, randomized study that will compare activity levels in patients who complete cardiac rehabilitation after clinically indicated percutaneous coronary intervention with and without use of the wrist-worn Fitbit Charge HR device and mobile platform application.

Primary Endpoint: The average number of steps taken per day will serve as the main marker of daily physical activity.

Control: Patients who do not receive the device (Fitbit Charge HR).

Secondary Endpoints: (1) change in daily energy expenditure (2) change in number of activity and sedentary bouts (3) change in sleep efficiency (4) change in weekly time of moderate/vigorous physical activity (5) change in quality of life (6) change in indicators of depression (7) change in medication adherence(8) change in HDL and LDL cholesterol (9) change in BMI and waist circumference (10) change in resting heart rate and blood pressure (11) change in exercise stress test performance (timeframe for all: baseline - 12 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Willing and able to give informed consent
* Successful, clinically-indicated PCI with no plan for staged procedure
* Clinically stable and able to exercise
* Access to smartphone (Apple or Android platform)
* Completed 10 weeks of CR and is expected to graduate program.

Exclusion Criteria:

* Plan for PCI or other major surgical procedure, which would limit exercise capability, within the 14 weeks following study enrollment.
* Home oxygen requirement
* Amputation, peripheral arterial disease, other musculoskeletal or neurological disease affecting mobility
* End-stage renal disease
* Ongoing Unstable angina or CCS IV angina
* NYHA IV heart failure
* Terminal illness
* Dementia
* Fall risk (inability to hold semi-tandem stance for 10 seconds)
* Pregnant women and prisoners
* Any other criteria that in the opinion of the investigator would preclude patient participation in the study and/or impact exercise capability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Relative change in average number of steps taken per day | Baseline and 12 weeks after completion of cardiac rehabilitation

SECONDARY OUTCOMES:
Relative change in average daily energy expenditure measured in % change in the average number of calories (kcal) expended per day | Baseline and 12 weeks after completion of cardiac rehabilitation
  Average daily energy expenditure will be measured in kcal/day by the Actigraph wGT3X-BT device.
Relative change in average number of daily activity bouts measured in % change in the average number of activity bouts per day | Baseline and 12 weeks after completion of cardiac rehabilitation
  Activity bouts will be measured as periods of continuous activity recorded by the Actigraph wGT3X-BT device.
Relative change in average number of daily sedentary bouts measured in % change in the average number of sedentary bouts per day | Baseline and 12 weeks after completion of cardiac rehabilitation
  Sedentary bouts will be measured as periods of prolonged inactivity recorded by the Actigraph wGT3X-BT device. Non-wear time periods are excluded from this analysis.
Relative change in average daily sleep efficiency measured in % change in average sleep efficiency. Sleep efficiency will also be measured in %. | Baseline and 12 weeks after completion of cardiac rehabilitation
  Sleep efficiency will be measured in % using data from the Actigraph wGT3X-BT device.
Relative change in average weekly moderate/vigorous physical activity, measured in % change in minutes spent in moderate/vigorous physical activity per week | Baseline and 12 weeks after completion of cardiac rehabilitation
  change in weekly time of moderate/vigorous physical activity (MVPA, defined as activity intensity of ≥3.0 metabolic equivalents [MET] or ≥100 steps/min) (minutes).
Relative change in quality of life, measured in % change in SF-36 health survey questionnaire score | Baseline and 12 weeks after completion of cardiac rehabilitation
  change in quality of life (as assessed by the Short Form Health (SF36) questionnaire).
Relative change in indicators of depression, measured in % change in PHQ9 questionnaire score | Baseline and 12 weeks after completion of cardiac rehabilitation
  change in indicators of depression (as assessed by the Patient Health (PHQ9) questionnaire).
Relative change in medication adherence, measured in % change in MMAS questionnaire score | Baseline and 12 weeks after completion of cardiac rehabilitation
  change in medication adherence (as assessed by the Morisky Medication Adherence Scale (MMAS-8).
Relative change in HDL and LDL cholesterol | Baseline and 12 weeks after completion of cardiac rehabilitation
Relative change in BMI | Baseline and 12 weeks after completion of cardiac rehabilitation
Relative change in resting heart rate | Baseline and 12 weeks after completion of cardiac rehabilitation
Relative change in exercise stress test performance | Baseline and 12 weeks after completion of cardiac rehabilitation
Relative change in blood pressure (BP) | Baseline and 12 weeks after completion of cardiac rehabilitation
Relative change in waist circumference | Baseline and 12 weeks after completion of cardiac rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Study Chair — North Texas Veterans Healthcare System

REFERENCES:
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. Circulation. 2011 Dec 6;124(23):e574-651. doi: 10.1161/CIR.0b013e31823ba622. Epub 2011 Nov 7. No abstract available. PMID 22064601
- [Background] Goel K, Lennon RJ, Tilbury RT, Squires RW, Thomas RJ. Impact of cardiac rehabilitation on mortality and cardiovascular events after percutaneous coronary intervention in the community. Circulation. 2011 May 31;123(21):2344-52. doi: 10.1161/CIRCULATIONAHA.110.983536. Epub 2011 May 16. PMID 21576654
- [Background] Moore SM, Dolansky MA, Ruland CM, Pashkow FJ, Blackburn GG. Predictors of women's exercise maintenance after cardiac rehabilitation. J Cardiopulm Rehabil. 2003 Jan-Feb;23(1):40-9. doi: 10.1097/00008483-200301000-00008. PMID 12576911
- [Background] Dolansky MA, Stepanczuk B, Charvat JM, Moore SM. Women's and men's exercise adherence after a cardiac event. Res Gerontol Nurs. 2010 Jan;3(1):30-8. doi: 10.3928/19404921-20090706-03. Epub 2010 Jan 27. PMID 20128541
- [Background] Moore SM, Charvat JM, Gordon NH, Pashkow F, Ribisl P, Roberts BL, Rocco M. Effects of a CHANGE intervention to increase exercise maintenance following cardiac events. Ann Behav Med. 2006 Feb;31(1):53-62. doi: 10.1207/s15324796abm3101_9. PMID 16472039
- [Background] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834
- [Background] Izawa KP, Watanabe S, Omiya K, Hirano Y, Oka K, Osada N, Iijima S. Effect of the self-monitoring approach on exercise maintenance during cardiac rehabilitation: a randomized, controlled trial. Am J Phys Med Rehabil. 2005 May;84(5):313-21. doi: 10.1097/01.phm.0000156901.95289.09. PMID 15829777
- [Background] Bohannon RW. Number of pedometer-assessed steps taken per day by adults: a descriptive meta-analysis. Phys Ther. 2007 Dec;87(12):1642-50. doi: 10.2522/ptj.20060037. Epub 2007 Oct 2. PMID 17911274
- [Background] VanWormer JJ, Boucher JL, Pronk NP, Thoennes JJ. Lifestyle behavior change and coronary artery disease: effectiveness of a telephone-based counseling program. J Nutr Educ Behav. 2004 Nov-Dec;36(6):333-4. doi: 10.1016/s1499-4046(06)60406-5. No abstract available. PMID 15617619